CLINICAL TRIAL: NCT01407978
Title: Tolerability and Immunogenicity Study of FLUVAL P H1N1 Monovalent Influenza Vaccine of Omninvest in Children and Adolescents
Brief Title: Tolerability and Immunogenicity Study of FLUVAL P H1N1 Flu Vaccine of Omninvest in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fluart Innovative Vaccine Ltd, Hungary (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLUVAL P-H-07
Record Dates: First submitted 2010-03-30; First posted 2011-08-02 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Novel 2009 Influenza H1N1; Influenza, Human
Keywords: Influenza; Pandemic vaccine; Seasonal vaccine; Prevention; Influenza vaccine; Influenza in humans; Pandemic influenza in humans; Influenza vaccine for children; Influenza vaccine for adolescents; Seasonal vaccine for children; Seasonal vaccine for adolescents
MeSH Terms: conditions — Influenza, Human | interventions — Vaccination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaccination with Fluval AB Novo (Active Comparator): * Vaccination with Fluval AB Novo trivalent influenza vaccine with 6 μg HA/0.5ml/strain active ingredient content and aluminium phosphate gel adjuvant.
  * Dose: 0.25 ml /total 3x3 μg HA/ in age group 3-12 years, 0.5 ml /total 3x6 μg HA/ in age group 12-18 years, single dose.
  Interventions: Biological: Vaccination with Fluval AB Novo
- Vaccination with Fluval AB (Active Comparator): * Vaccination with Fluval AB trivalent influenza vaccine with 15 μg HA/0.5ml/strain active ingredient content and aluminium phosphate gel adjuvant.
  * Dose: 0.25 ml /total 3x7.5 μg HA/ in age group 3-12 years, 0.5 ml /total 3x15 μg HA/ in age group 12-18 years, single dose.
  Interventions: Biological: Vaccination with Fluval AB
- Vaccination with Fluval P (Experimental): * Vaccination with Fluval P monovalent influenza vaccine with 6 μg HA/0.5 ml active ingredient content and aluminium phosphate gel adjuvant.
  * Dose: 0.25 ml /total 3 μg HA/ in age group 3-12 years, and 0.5 ml /total 6 μg HA/ in age group 12-18 years, single dose.
  Interventions: Biological: Vaccination with Fluval P monovalent influenza vaccine

INTERVENTIONS:
Biological: Vaccination with Fluval P monovalent influenza vaccine — * Vaccination with Fluval P monovalent influenza vaccine with 6 μg HA/0.5 ml active ingredient content and aluminium phosphate gel adjuvant.
  * Dose: 0.25 ml /total 3 μg HA/ in age group 3-12 years, and 0.5 ml /total 6 μg HA/ in age group 12-18 years, single dose.
  Other Names: Fluval P; FL-P-K-01/09
  Arms: Vaccination with Fluval P
Biological: Vaccination with Fluval AB — * Vaccination with Fluval AB trivalent influenza vaccine with 15 μg HA/0.5ml/strain active ingredient content and aluminium phosphate gel adjuvant.
  * Dose: 0.25 ml /total 3x7.5 μg HA/ in age group 3-12 years, 0.5 ml /total 3x15 μg HA/ in age group 12-18 years, single dose.
  Other Names: Fluval AB; 5609
  Arms: Vaccination with Fluval AB
Biological: Vaccination with Fluval AB Novo — * Vaccination with Fluval AB Novo trivalent influenza vaccine with 6 μg HA/0.5ml/strain active ingredient content and aluminium phosphate gel adjuvant.
  * Dose: 0.25 ml /total 3x3 μg HA/ in age group 3-12 years, 0.5 ml /total 3x6 μg HA/ in age group 12-18 years, single dose.
  Other Names: Fluval AB Novo; FL-K-13/09
  Arms: Vaccination with Fluval AB Novo

SUMMARY:
This is a single-blind, reference drug controlled study to assess safety and tolerability of FLUVAL P H1N1 monovalent influenza vaccine (whole virus, inactivated, adjuvanted with alumn phosphate gel) containing 6 mcgHA per 0.5mL active ingredient in children and adolescents. To assess, as secondary objective, the efficacy (immunogenicity) of the vaccine by serology testing.

DETAILED DESCRIPTION:
Primary Objective:

* To assess tolerability/safety (incidence of adverse events 21-28 days following vaccination) of the study drug.

Secondary Objectives:

* To assess the efficacy (immunogenicity) of the study drug by serology testing of blood samples taken at Day 21-28 after immunization in groups and age groups.
* To assess long term (180-210 days following vaccination) tolerability/safety (incidence of adverse events) of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 12 years, adolescents aged 12 to 18 years, both sexes;
* Are in good health (as determined by vital signs and existing medical condition) or are in stable medical condition. Subjects will not be excluded with known adequately treated clinically significant organ or systemic diseases (e.g. asthma or diabetes)m such that, in the opinion of the investigator, the significance of the disease will not compromise the subject's participation in the study.
* Female volunteers of childbearing potential with a negative result from the urine pregnancy test prior to vaccination who agrees to use an acceptable contraception method (includes implants, injectibles, combined oral contraceptives, effective intrauterine devices /IUDs/, sexual abstinence, or a vasectomized partner) or abstinence throughout the trial and not become pregnant for the duration of the study.
* Capability of adolescent participants aged 12 to 18 years and the legitimate representative of all volunteers to understand and comply with planned study procedures;
* Absence of existence of any exclusion criteria.

Exclusion Criteria:

* Pregnancy or breast feeding or positive urine pregnancy test at baseline prior to vaccination;
* Known allergy to eggs or other components of the vaccine (in particular mercury);
* History of Guillain-Barré syndrome;
* Active neoplasm (i.e. requiring any form of anti-neoplastic therapy);
* Immunosuppressive therapy in the preceding 36 months;
* Concomitant corticosteroid therapy, including high-dose inhaled corticosteroids (local corticosteroid or corticosteroid nasal spray are permitted);
* Immunoglobulin (or similar blood product) therapy within 3 months prior to vaccination;
* Documented HIV, HBV or HCV infection;
* Chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the immunoresponse;
* Acute febrile respiratory illness within one week prior to vaccination;
* Vaccine therapy within 4 weeks prior to vaccination;
* Influenza vaccination within 6 months prior to vaccination;
* Experimental drug therapy within 1 month prior to vaccination;
* Past or current psychiatric disease of the volunteer or the legitimate representative that upon judgement of the investigator may have effect on the objective decision-making of the volunteer or the legitimate representative;
* Alcohol or drug abuse of the participant or the legitimate representative.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 21-28 days after vaccination

SECONDARY OUTCOMES:
Post vaccination HI antibody titer | 21-28 days after vaccination
Incidence of adverse events | 180-210 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ősi, Dr., Study Director — Omninvest Ltd.; Éva Szabó, MD, Principal Investigator — "Csolnoky Ferenc" Veszprém County Hospital
Locations (1):
- "Csolnoky Ferenc" Veszprém County Hospital, Veszprém, Veszprém megye, Hungary